CLINICAL TRIAL: NCT05364086
Title: Disparities in Results of Immune Checkpoint Inhibitor Treatment (DiRECT): A Prospective Cohort Study of Cancer Survivors Treated With Anti-PD-1/Anti-PD-L1 Immunotherapy in a Community Oncology Setting
Brief Title: An Observational Research Study for Cancer Patients on Immune Checkpoint Inhibitors, DiRECT Study
Acronym: DiRECT
Status: Recruiting | Type: Observational
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Charles Kamen, URCC Study Chair, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Other Study IDs: URCC21038; NCI-2022-01426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC21038 (Other: University of Rochester NCORP Research Base); URCC-21038 (Other: DCP); URCC-21038 (Other: CTEP); UG1CA189961 (NIH); UH3CA260602 (NIH)
Record Dates: First submitted 2022-03-31; First posted 2022-05-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Specimen Handling; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor, blood, saliva and stool
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaire, biospecimen, medical records)): Patients complete questionnaires and undergo collection of blood, saliva and optional stool samples before 1st and 2nd infusion of immunotherapy. Patients also complete additional questionnaires undergo additional collection of blood samples 6 months after 1st infusion of immunotherapy and then every year after 1st infusion of immunotherapy. A tumor sample will also be collected at the beginning of the study and patients medical records will be reviewed. Patients may also optionally complete an interview following their 2nd infusion of immunotherapy.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tumor, blood, saliva and stool samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Review of medical records
Other: Interview — Complete an interview
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study compares treatment outcomes between patients of African American/Black (AA) ancestry and European American/White (EA) ancestry currently receiving immune checkpoint inhibitor treatment. Collecting samples of blood and saliva and health and treatment information from racially diverse patients receiving immune checkpoint inhibitor treatment over time may help doctors better understand health care disparities among all cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare incidence of Common Terminology Criteria for Adverse Events (CTCAE) grade 2-5 immune-related adverse reactions (irAEs) between African American (AA) and European American (EA) patients within the first year of starting immune checkpoint inhibitor (ICI) treatment.

SECONDARY OBJECTIVES:

I. To compare objective response rate (ORR) to ICI treatment between AA and EA patients within the first year of starting ICI treatment.

II. To compare health-related quality of life (HRQOL) measured using the Patient Reported Outcomes Measurement Information System (PROMIS) Preference (Patient Reported Outcomes [PRO] Pr) summary score and Functional Assessment of Cancer Therapy-Immune Checkpoint Modulator (FACT-ICM) between AA and EA patients within 1 year of starting ICI treatment.

EXPLORATORY OBJECTIVES:

I. To compare AA and EA patients on severity (i.e., CTCAE grade) and timing of irAEs within 1 year of starting ICI treatment.

II. To assess disease, treatment, individual, and behavioral factors as predictors of grade 2-5 irAEs, and as potential causes of racial differences in irAEs, within 1 year of starting ICI treatment.

III. To compare AA and EA patients on long-term outcomes (e.g., progression-free survival [PFS], overall survival [OS], and HRQOL beyond the first year) at the end of the study period.

IV. To assess the impact of irAEs and disease, treatment, behavioral, and individual factors on ICI outcomes (ORR, HRQOL, PFS, OS), and as potential causes of racial differences in outcomes, at the end of the study period.

V. To compare ICI treatment patterns (e.g., delay and discontinuation of ICI treatment) between AA and EA patients within 1 year of starting ICI treatment.

VI. To assess irAEs, treatment, disease, and individual factors, including healthcare barriers, as possible reasons for suboptimal treatment patterns, and as potential causes of racial differences, within 1 year of starting ICI treatment.

VII. To collect optional stool samples and an additional blood sample at the time of the occurrence of grade 3-4 irAEs to strengthen the biobank for future research on ICI response and racial disparities.

OUTLINE: This is an observational study.

Patients complete questionnaires and undergo collection of blood, saliva, and optional stool samples before 1st and 2nd infusion of immunotherapy. Patients also complete additional questionnaires undergo additional collection of blood samples 6 months after 1st infusion of immunotherapy and then every year after 1st infusion of immunotherapy. A tumor sample will also be collected at the beginning of the study and patients medical records will be reviewed. Patients may also optionally complete an interview following their 2nd infusion of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Self-identify as African/African American/black (AA), or European American/ Caucasian/white (EA)

  * Patients may identify a Hispanic/Latino ethnicity in combination with an AA or EA racial identity
* Have a current diagnosis of invasive cancer at stage I-IV

  * Patients may have a history of previous cancer diagnosis and cancer treatment not involving immunotherapy
* Be scheduled to receive anti-PD-1/-L1 ICI-containing therapy alone or in combination with co-treatments (including alternative ICIs)
* Be able to speak and read English or Spanish
* Be able to provide informed consent

Exclusion Criteria:

* Identify as Asian, Pacific Islander, or American Indian/Alaskan Native
* Be diagnosed with melanoma (because melanoma is very rare in AAs)
* Currently participate in any trials of a cancer therapeutic nature; participation in noninterventional trial, or trials of symptom control or supportive nature is allowed; participation in future cancer therapeutic trials after completing the A2 assessment (e.g., after the second infusion of ICIs) is also allowed
* Have received prior immunotherapy for cancer, including checkpoint inhibitors, chimeric antigen receptor (CAR)-T therapy, cytokine therapy, and/or Bacillus Calmette-Guerin (BCG) for bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African American or European American patients diagnosed with stage I-IV invasive cancer receiving immune checkpoint inhibitor treatment
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Racial differences in the incidence of Common Terminology Criteria for Adverse Events (CTCAE) grade 2-5 immune-related adverse reactions (irAEs) | Within 1 year after starting immune checkpoint inhibitor (ICI) treatment
  Will be evaluated in bivariate analysis by Chi-square, Wilcoxon rank-sum test, or two sample t-tests.

SECONDARY OUTCOMES:
Racial differences in overall response rate (ORR) between African American (AA) and European American (EA) patients | Within 1 year after starting ICI treatment
  Multivariable modeling will be conducted to adjust for covariates.
Health-related quality of life (HRQOL) - PROPr | Within 1 year after starting ICI treatment
  Will be assessed by Patient Reported Outcomes Preference (PROPr). This is a T-score with a mean of 50 and a standard deviation of 0.
Health-related quality of life (HRQOL) - FACT-ICM | Within 1 year after starting ICI treatment
  Will be assessed by Functional Assessment of Cancer Therapy-Immune Checkpoint Modulator (FACT-ICM), which is a count of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kamen, PhD, Principal Investigator — University of Rochester NCORP Research Base
Locations (259):
- United States (259):
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Tift Regional Medical Center, Tifton, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - MBP Cancer Center - Baton Rouge General, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Cancer Center of Acadiana, Lafayette, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Jackson Oncology Associates PLLC, Jackson, Mississippi
  - Mississippi Baptist Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Waccamaw Oncology - Georgetown, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Waccamaw Oncology-Murrells Inlet, Murrells Inlet, South Carolina
  - Waccamaw Oncology-Myrtle Beach, Myrtle Beach, South Carolina
  - Beaufort Memorial/New River Cancer Center, Okatie, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Valley Medical Center, Renton, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin